CLINICAL TRIAL: NCT00363675
Title: Evaluation of Hand Assessments in Children With Severe Hand Burns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This was a pilot study, but the larger study was not funded.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Mary Jo Baryza, Director of Therapeutic Services, Shriners Hospitals for Children, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-P000388/3
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Results first posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-02

CONDITIONS: Burns
Keywords: Hand Burns; Pediatrics
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All study participants (Experimental): Children with hand burns
  Interventions: Behavioral: Functional hand tests

INTERVENTIONS:
Behavioral: Functional hand tests — Chilren were tested after healed hand burns for functional ability.

SUMMARY:
This study is designed to see if some tests of hand movement, strength, and function are valid for children with burns.

DETAILED DESCRIPTION:
Children will be given a battery of tests to determine the validity of these measures for children with severe hand burns. The tests include:

* Pinch and grip strength;
* Stereognosis;
* Speed of manipulation using the Nine Hole Peg Test, Box & Blocks Test, and the Moberg Pickup Test;
* Measurement of Range of Motion of the wrist and fingers.

ELIGIBILITY:
Inclusion Criteria:

* Third degree brns to one or both hands
* All areas closed
* Age between 5 and 18 years old
* English or Spanish speaking

Exclusion Criteria:

* Previous hand condition
* Unable to follow 2 step directions

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2006-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jo Baryza, MS, PT, PCS, Principal Investigator — Shriners Hospitals for Children - Boston
Locations (1):
- Shriners Hospitals for Children - Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Children were administered hand assessments to measure function after hand burns by a trained therapist.
Period: Overall Study
Arm/Group | All Study Participants
Started | 3
Completed Testing | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Blocks & Box (Standardized Test).
Description: Children are asked to move as many blocks as possible from one box to another in one minute. The number of blocks moved is the score.
Time Frame: Baseline
Population: Convenience sample was planned for this study.
Measure: Median (Full Range); unit: Blocks
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Blocks | 32 [21 to 37]

2. Primary Outcome: Range of Motion, Total Active Motion (TAM)
Description: Subjects' degrees of hand motion are measured by a trained therapist and recorded. Total Active Motion is a measure of finger range of motion that can be used to predict functional movement of the hand. The TAM is the sum of the degrees of active motion of each of the three joints of the fingers, and two joints of the thumb. For this study we also included wrist motion. Full TAM is 1,455 degrees of motion.
Time Frame: Baseline
Population: Convenience sample was planned for ths study.
Measure: Median (Full Range); unit: Degrees
Groups:
- Normal as Defined by Hand Therapist.: Children were administered hand assessments to measure function after hand burns by a trained therapist.
Arm/Group | Normal as Defined by Hand Therapist.
Number analyzed (Participants) | 3
Degrees | 998 [901 to 1260]

3. Primary Outcome: Grip Strength
Description: This is a measure of grip strength in pounds using a dynamometer. The subject squeezes the dynamometer as hard as possible for three trials separated by a short rest. The mean of the three trials is the score.
Time Frame: Baseline
Population: Convenience sample was planned for this study.
Measure: Median (Full Range); unit: Pounds
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Pounds | 7.33 [4 to 9.17]

4. Primary Outcome: Moberg Pickup Test
Description: The child picks up 12 small objects such as a coin, safety pin and paper clip one at a time and puts them in a container. The time in seconds to complete the task is the score.
Time Frame: Seconds to pick up all 12 objects
Population: A convenience sample was planned for this study.
Measure: Median (Full Range); unit: Seconds
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Seconds | 19 [16 to 48]

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
This pilot study was discontinued secondary to lack of grant funding for the project.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes